CLINICAL TRIAL: NCT01748513
Title: Morbid Obesity and Optimization of Preoperative Fluid Therapy
Brief Title: Volume-challenge in Morbid Obesity
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tomi Pösö, MD, Umeå University
Other Study IDs: 09-042M
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Anomaly; Venous Return
Keywords: morbidly obese patients,; preoperative volume-challenge,; transthoracic echocardiography,; TTE,; rapid weight loss,; venous return,; bariatric surgery,; left ventricular outflow tract,; stroke volume,; diastolic function,; hypervolemia,; hypovolemia
MeSH Terms: conditions — Congenital Abnormalities; Edema; Hypovolemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- preoperative venous return optimizing: Morbidly obese patients scheduled for bariatric surgery
  Interventions: Other: preoperative venous return optimizing

INTERVENTIONS:
Other: preoperative venous return optimizing — Preoperative transthoracic echocardiography (TTE) was performed in the awake state before and after volume challenge based on 6ml colloids /kg ideal body weight.

SUMMARY:
Preoperative venous return stability and euvolemia is essential in management of morbidly obese patients. Fluid therapy regimes for patients with high BMI, especially with focus on preoperative management, are rare and not in consensus.The aim of this study was to evaluate preoperative effects of a standardized, ideal body weight (IBW) based volume-challenge on hemodynamics, stroke volume and level of venous return to the heart.

DETAILED DESCRIPTION:
34 morbidly obese patients scheduled for bariatric surgery underwent a preoperative three-week preparation by rapid-weight-loss-diet (RWL) to be accepted for bariatric surgery. Preoperative transthoracic echocardiography (TTE) was performed in the awake state before and after volume-challenge (VC) based on 6ml colloids /kg IBW. Feasibility of standardized VC was evaluated by TTE. Dynamic and non-dynamic echocardiographic indices for VC were studied.

Main outcome measures: Volume-responsiveness and level of venous return before and after volume-challenge were assessed by TTE. An increase of stroke volume ≥ 13% was considered as a volume-responder.

ELIGIBILITY:
Inclusion Criteria:

* enrolled for bariatric surgery
* BMI ≥ 40 or ≥ 35kg/m2 with co-morbidities
* preoperative three-weeks preparation by rapid-weight-loss-diet and weight loss

Exclusion Criteria:

* untreated significant hypertension
* unstable angina pectoris
* significant valve regurgitation or stenosis
* known severe pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients scheduled for bariatric surgery in Northern part of Sweden; Norrbotten county council.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
level of venous return | 0,1 hour

SECONDARY OUTCOMES:
Volume-responsiveness | 0,1 hour

OTHER OUTCOMES:
Evaluation of feasibility of dynamic and non-dynamic echocardiographic indices for volume challenge | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Tomi P Pösö, MD, Principal Investigator — Norrbotten county council, Umeå University
Locations (1):
- Sunderby county hospital, Luleå, Norrbotten County, Sweden